CLINICAL TRIAL: NCT02037698
Title: Role of CT Scan for the Successful Recanalization of Chronic Total Occlusion; a Randomized Comparison Between 3D CT-guided PCI vs. Conventional Treatment (CT-CTO Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2013-0062
Record Dates: First submitted 2013-12-18; First posted 2014-01-16 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Obstructive Disease; Chronic Total Occlusion Lesions
Keywords: CTO; CT; Revascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-PCI CT scan group (Experimental): Pre-PCI CT scan
  Interventions: Device: Pre-PCI coronary CT scan
- Control group (No Intervention): Control

INTERVENTIONS:
Device: Pre-PCI coronary CT scan — Coronary CT scan before CTO PCI
  Arms: Pre-PCI CT scan group

SUMMARY:
The revascularization of chronic total occlusion of coronary arteries (CTO) is the most challenging procedure for the coronary intervention. For the initial period for CTO intervention, percutaneous coronary artery intervention (PCI) of CTO lesions are associated with low procedural success rates about 70%. Recently, the success rate of the recanalization of CTOs has been raised in several studies.

Coronary CT angiography (CCTA) is an effective noninvasive diagnostic modality for detecting coronary artery disease. CCTA can visualize the complete anatomy of coronary arteries in contrast to conventional coronary angiography, reducing the deferral rates from CTO intervention. Assessment of characteristics of CTO lesions by pre-procedural CCTA could help to determine revascularization strategy and estimate the procedure time, leading to lower procedural complications. We suggest that success rates and clinical outcome of intervention of CTO lesion can be improved by pre-procedural CCTA.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age >19 years) with CTO (TIMI = 0 and estimated duration of occlusion at least 3 months)
* Typical symptomatic angina or positive stress test in various functional studies evaluating ischemia
* Eligible patients for pre-procedural CT scan and coronary angiogram

Exclusion Criteria:

* Cardiogenic shock or ejection fraction < 25%
* CTO lesions at DES restenosis or graft occlusion lesion
* Significant left main stenosis
* Retry of same CTO lesion within 2 weeks
* Acute myocardial infarction within 48 hours
* Hypersensitivity to aspirin, clopidogrel, or -limus families / or contraindication to antiplatelet agents
* Severe hepatic dysfunction (≥3 times normal reference values)
* Life expectancy < 1 years
* Pregnant women or women with potential childbearing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Successful CTO recanalization | Immediately after CTO PCI
  Incidence of the successful CTO recanalization between pre-PCI CT scan group versus control group

SECONDARY OUTCOMES:
Incidence of MACEs | 12 months after index PCI
  Comparison of major adverse cardiac events (MACE), between ZES and EES implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Hong SJ, Kim BK, Cho I, Kim HY, Rha SW, Lee SH, Park SM, Kim YH, Chang HJ, Ahn CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y; CT-CTO Investigators. Effect of Coronary CTA on Chronic Total Occlusion Percutaneous Coronary Intervention: A Randomized Trial. JACC Cardiovasc Imaging. 2021 Oct;14(10):1993-2004. doi: 10.1016/j.jcmg.2021.04.013. Epub 2021 Jun 16. PMID 34147439